CLINICAL TRIAL: NCT06926062
Title: Implementing a Proactive Approach to Communicate and Teach About HPV Vaccination in Pharmacies: IMPACT HPV Study
Brief Title: Interpersonal Communication Training and Vaccination Workflow Training Alone and in Combination to Improve Communication and Recommendations About HPV Vaccination in Pharmacies, IMPACT HPV Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Health Services Research
Other Study IDs: RG1125096; NCI-2025-01610 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 20694 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2025-03-19; First posted 2025-04-13 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-07

CONDITIONS: Human Papillomavirus-Related Carcinoma
MeSH Terms: interventions — Practice Guidelines as Topic; Standard of Care; Early Intervention, Educational; Educational Status; Methods; Interviews as Topic; Vaccination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (10):
- Objective 1, Topic I (safety and side effects survey) (Other): Parents review 4 messages on safety and side effects and complete a survey over 15-20 minutes in support of intervention refinement on study.
  Interventions: Other: Educational Intervention; Other: Questionnaire Administration
- Objective 1, Topic II (vaccine effectiveness survey) (Other): Parents review 4 messages on vaccine effectiveness and complete a survey over 15-20 minutes in support of intervention refinement on study.
  Interventions: Other: Educational Intervention; Other: Questionnaire Administration
- Objective 1, Topic III (sexual activity survey) (Other): Parents review 4 messages on sexual activity and complete a survey over 15-20 minutes in support of intervention refinement on study.
  Interventions: Other: Educational Intervention; Other: Questionnaire Administration
- Objective 1, Topic IV (HPV vaccine for boys survey) (Other): Parents review 4 messages on HPV vaccine for boys and complete a survey over 15-20 minutes in support of intervention refinement on study.
  Interventions: Other: Educational Intervention; Other: Questionnaire Administration
- Objective 1, Topic V (age to start vaccine survey) (Other): Parents review 4 messages on age to start vaccine and complete a survey over 15-20 minutes in support of intervention refinement on study.
  Interventions: Other: Educational Intervention; Other: Questionnaire Administration
- Objective 1, Topic VI (school entry requirements survey) (Other): Parents review 4 messages on school entry requirements and complete a survey over 15-20 minutes in support of intervention refinement on study.
  Interventions: Other: Educational Intervention; Other: Questionnaire Administration
- Objective 2, Group I (control) (Active Comparator): Pharmacy staff provide vaccinations per usual care.
  Interventions: Other: Best Practice; Other: Interview; Other: Questionnaire Administration
- Objective 2, Group II (strategy A) (Experimental): Pharmacy staff receive interpersonal communication training over 120 minutes and provide vaccinations using the interpersonal communication strategy.
  Interventions: Other: Interview; Other: Questionnaire Administration; Behavioral: Training and Education; Procedure: Vaccination
- Objective 2, Group III (strategy B) (Experimental): Pharmacy staff receive the vaccination workflow training and provide vaccinations using the vaccination workflow training strategy.
  Interventions: Other: Interview; Other: Questionnaire Administration; Behavioral: Training and Education; Procedure: Vaccination
- Objective 2, Group IV (strategies A and B) (Experimental): Pharmacy staff receive interpersonal communication training as well as vaccination workflow training and provide vaccinations using both the interpersonal communication strategy and the vaccination workflow training strategy.
  Interventions: Other: Interview; Other: Questionnaire Administration; Behavioral: Training and Education; Procedure: Vaccination

INTERVENTIONS:
Other: Best Practice — Provide vaccinations per usual care
  Other Names: standard of care; standard therapy
  Arms: Objective 2, Group I (control)
Other: Educational Intervention — Review messages on safety and side effects
  Other Names: Education for Intervention; Intervention by Education; Intervention through Education; Intervention, Educational
  Arms: Objective 1, Topic I (safety and side effects survey)
Other: Educational Intervention — Review messages on vaccine effectiveness
  Other Names: Education for Intervention; Intervention by Education; Intervention through Education; Intervention, Educational
  Arms: Objective 1, Topic II (vaccine effectiveness survey)
Other: Educational Intervention — Review messages on sexual activity
  Other Names: Education for Intervention; Intervention by Education; Intervention through Education; Intervention, Educational
  Arms: Objective 1, Topic III (sexual activity survey)
Other: Educational Intervention — Review messages on HPV vaccine for boys
  Other Names: Education for Intervention; Intervention by Education; Intervention through Education; Intervention, Educational
  Arms: Objective 1, Topic IV (HPV vaccine for boys survey)
Other: Educational Intervention — Review message on age to start vaccine
  Other Names: Education for Intervention; Intervention by Education; Intervention through Education; Intervention, Educational
  Arms: Objective 1, Topic V (age to start vaccine survey)
Other: Educational Intervention — Review messages on school entry requirements
  Other Names: Education for Intervention; Intervention by Education; Intervention through Education; Intervention, Educational
  Arms: Objective 1, Topic VI (school entry requirements survey)
Other: Interview — Ancillary studies
  Arms: Objective 2, Group I (control); Objective 2, Group II (strategy A); Objective 2, Group III (strategy B); Objective 2, Group IV (strategies A and B)
Other: Questionnaire Administration — Complete a survey
  Arms: Objective 1, Topic I (safety and side effects survey); Objective 1, Topic II (vaccine effectiveness survey); Objective 1, Topic III (sexual activity survey); Objective 1, Topic IV (HPV vaccine for boys survey); Objective 1, Topic V (age to start vaccine survey); Objective 1, Topic VI (school entry requirements survey)
Other: Questionnaire Administration — Ancillary studies
  Arms: Objective 2, Group I (control); Objective 2, Group II (strategy A); Objective 2, Group III (strategy B); Objective 2, Group IV (strategies A and B)
Behavioral: Training and Education — Receive interpersonal communication training
  Arms: Objective 2, Group II (strategy A); Objective 2, Group IV (strategies A and B)
Behavioral: Training and Education — Receive the vaccination workflow training
  Arms: Objective 2, Group III (strategy B); Objective 2, Group IV (strategies A and B)
Procedure: Vaccination — Provide vaccinations using the interpersonal communication strategy
  Arms: Objective 2, Group II (strategy A)
Procedure: Vaccination — Provide vaccinations using the vaccination workflow training strategy
  Arms: Objective 2, Group III (strategy B)
Procedure: Vaccination — Provide vaccinations using both the interpersonal communication strategy and the vaccination workflow training strategy
  Arms: Objective 2, Group IV (strategies A and B)

SUMMARY:
This clinical trial compares usual care to interpersonal communication training and vaccination workflow training, alone or in combination, for improving communication about and recommendations for human papillomavirus (HPV) and other vaccinations in pharmacies. Low HPV vaccination in the United States has placed unvaccinated children at risk of developing cancers as adults that could have been prevented. Pharmacies can be convenient for vaccination because they are open longer hours, have shorter wait times, can see patients without appointments and may cost less. However, many people are not aware that vaccination is available in pharmacies and some pharmacies lack the commitment from staff to vaccinate or may not have protocols in place for vaccination. Proactive communication approaches to recommending HPV vaccination have been shown to be effective in medical offices but have not been tested in the pharmacy setting. Interpersonal communication training incorporates the 5 A's (assess, advice, agree, assist and arrange) behavioral counseling framework to strongly recommend HPV and other vaccines and effectively answer any questions or concerns about vaccination. Vaccination workflow training establishes vaccination decision support strategies that pharmacies use to improve vaccination workflows. Interpersonal communication training and vaccination workflow training alone or in combination may improve communication and recommendations for HPV vaccination and increase HPV vaccination in pharmacies.

DETAILED DESCRIPTION:
OUTLINE:

OBJECTIVE 1: Parents are randomized to receive messages on 1 of 6 topics.

TOPIC I (SAFETY AND SIDE EFFECTS): Parents review 4 messages on safety and side effects and complete a survey over 15-20 minutes in support of intervention refinement on study.

TOPIC II (VACCINE EFFECTIVENESS): Parents review 4 messages on vaccine effectiveness and complete a survey over 15-20 minutes in support of intervention refinement on study.

TOPIC III (SEXUAL ACTIVITY): Parents review 4 messages on sexual activity and complete a survey over 15-20 minutes in support of intervention refinement on study.

TOPIC IV (HPV VACCINE FOR BOYS): Parents review 4 messages on HPV vaccine for boys and complete a survey over 15-20 minutes in support of intervention refinement on study.

TOPIC V (AGE TO START VACCINE): Parents review 4 messages on age to start vaccine and complete a survey over 15-20 minutes in support of intervention refinement on study.

TOPIC VI (SCHOOL ENTRY REQUIREMENTS): Parents review 4 messages on school entry requirements and complete a survey over 15-20 minutes in support of intervention refinement on study.

OBJECTIVE 2: Pharmacies are assigned to a strata of 4 pharmacies with similar characteristics and pharmacies within each strata are randomized to 1 of 4 groups.

GROUP I (CONTROL): Pharmacy staff provide vaccinations per usual care.

GROUP II (STRATEGY A): Pharmacy staff receive interpersonal communication training over 120 minutes and provide vaccinations using the interpersonal communication strategy.

GROUP III (STRATEGY B): Pharmacy staff receive the vaccination workflow training and provide vaccinations using the vaccination workflow training strategy.

GROUP IV (STRATEGIES A AND B): Pharmacy staff receive interpersonal communication training as well as vaccination workflow training and provide vaccinations using both the interpersonal communication strategy and the vaccination workflow training strategy.

ELIGIBILITY:
Inclusion Criteria:

* OBJECTIVE 1: Adults aged 18 years or older who live in the 50 United States (U.S.) states and Washington District of Columbia (D.C.) and are parents or guardians of children ages 9-17 are eligible to take the national survey (n ≤ 1,600, with anticipated enrollment of n = ~1,500)
* OBJECTIVE 2: Pharmacy staff at participating pharmacies (n ≤ 100)
* OBJECTIVE 2: Adults aged 18 years or older whose children ages 9-17 received an HPV vaccine at one of the participating pharmacies in study year 2 (n ≤ 200)

Exclusion Criteria:

* OBJECTIVE 1: Non-English speaking as the survey is only available for this project in English
* OBJECTIVE 1: Parents whose index children have completed the HPV vaccine series
* OBJECTIVE 2: Non-English speaking as the study funding only provided resources for surveys and interview materials to be available in English
* OBJECTIVE 2: Parents whose index children have completed the HPV vaccine series

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1900 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Perceived fit, relevance, or compatibility of human papillomavirus (HPV) vaccination or the communication strategy for a given practice site, provider, or patient (Appropriateness: Pharmacy Staff) | At baseline, 2 months post-training delivery, and 12 months post-training delivery
  Assessed via survey. The survey was developed by study researchers based upon the Implementation Outcomes Questionnaire (IOQ) (Livet M, et al. 2021.). It was used to capture change of participants' perceptions pre/post training. There are five answers to each survey question and each answer is given a score from 1 to 5, with 1 being strongly disagree and 5 being strongly agree. Higher numerical scores on the 5-point scale indicate greater level of agreement that the intervention was appropriate to support HPV vaccination delivery to children ages 9-17. Study researchers will calculate the average scale based on numeric scores. For questions that are asked in a reverse fashion, study researchers will reverse the score accordingly.
Perceived fit, relevance, or compatibility of human papillomavirus (HPV) vaccination or the communication strategy for a given practice site, provider, or patient (Appropriateness: Parents) | The outcome will be measured at one time point, at a time frame from the date of vaccine administration to up to 8 weeks after that vaccine administration date
  Appropriateness outcomes will be assessed via survey to parents following their child's HPV vaccination. The four questions to evaluate appropriateness are sourced from evidence-based assessments of Intervention Appropriateness Measure (IAM) from Weiner et al. (2017). There are five answers to each survey question and each answer is given a score from 1 to 5, with 1 being strongly disagree and 5 being strongly agree. Higher numerical scores on the 5-point Likert scale indicate greater level of agreement that the intervention was appropriate in supporting HPV vaccination delivery to children ages 9-17.
Perceptions that HPV vaccinations or the communication strategy is agreeable, palatable, or satisfactory (Acceptability: Pharmacy Staff) | At baseline, 2 months post-training delivery, and 12 months post-training delivery
  Assessed via survey. The survey was developed by study researchers based upon the Implementation Outcomes Questionnaire (IOQ) (Livet M, et al. 2021.). It was used to capture change of participants' perceptions pre/post training. There are five answers to each survey question and each answer is given a score from 1 to 5, with 1 being strongly disagree and 5 being strongly agree. Higher numerical scores on the 5-point Likert scale indicate greater level of agreement that the intervention was acceptable to support HPV vaccination delivery to children ages 9-17. Study researchers will calculate the average scale based on numeric scores. For questions that are asked in a reverse fashion, study researchers will reverse the score accordingly.
Perceptions that HPV vaccinations or the communication strategy is agreeable, palatable, or satisfactory (Acceptability: Parents) | The outcome will be measured at one time point, at a time frame from the date of vaccine administration to up to 8 weeks after that vaccine administration date
  Acceptability outcomes will be assessed via survey to parents following their child's HPV vaccination. The four questions to evaluate acceptability are sourced from evidence-based assessments of Acceptability of Intervention Measure (AIM) from Weiner et al. (2017). There are five answers to each survey question and each answer is given a score from 1 to 5, with 1 being strongly disagree and 5 being strongly agree. Higher numerical scores on the 5-point Likert scale indicate greater level of agreement that the intervention was acceptable to support HPV vaccination delivery to children ages 9-17.
Extent to which the communication strategy was successfully implemented and used at pharmacies to support HPV vaccine delivery (Feasibility) | At baseline, 2 months post-training delivery, and 12 months post-training delivery
  Assessed via survey. The survey was developed by study researchers based upon the Implementation Outcomes Questionnaire (IOQ) (Livet M, et al. 2021.). It was used to capture change of participants' perceptions pre/post training. There are five answers to each survey question and each answer is given a score from 1 to 5, with 1 being strongly disagree and 5 being strongly agree. Higher numerical scores on the 5-point scale indicate greater level of agreement that the intervention was feasible to support HPV vaccination delivery to children ages 9-17. Study researchers will calculate the average scale based on numeric scores. For questions that are asked in a reverse fashion, study researchers will reverse the score accordingly.
HPV vaccination delivery (Fidelity: Pharmacy Staff) | Up to completion of the 12 month trial period
  Will conduct audits of the pharmacy electronic records to assess adherence to HPV vaccination protocols, by comparing the proportion of HPV vaccines given "on time" to children aged 9-10 and 11-12 versus "late" to children aged 13-17.
HPV vaccination delivery (Fidelity: Parents) | The outcome will be measured at one time point, at a time frame from the date of vaccine administration to up to 8 weeks after that vaccine administration date
  HPV vaccine delivery fidelity will be assessed via survey to parents following their child's HPV vaccination. Parents will be asked to indicate which of seven, if any, supportive vaccination behaviors occurred during their visit in a "select all that apply" format. The seven experiences correspond to vaccination behaviors that have been shown in formative research to support HPV vaccine delivery and parents' perceptions of acceptability and appropriateness of HPV vaccination workflows using the 5As Behavioral Counseling Model (Sturgiss et al. 2017). The supportive behaviors include eligibility screening, recommendation, counseling, documentation and record retrieval support, PCP reporting, and scheduling for follow up. To summarize the overall fidelity to the workflow per respondent, study researchers will create a composite "fidelity score" by summing the number of behaviors each parent endorsed (range: 0-7). Higher scores will indicate greater adherence to the recommended workflow.
Self-efficacy | At baseline, 2 months post-training delivery, and 12 months post-training delivery
  Assessed via survey. The survey was developed by study researchers and includes validated measures from a 31-item medication therapy management (MTM) efficacy scale (Martin B, et al. 2010) and a statewide survey of healthcare providers (McRee AL, et.al. 2014). It will be used to capture change of participants' perceptions pre/post training. For this outcome there are five answers to each survey question reflecting how confident the respondent is in performing tasks related to providing HPV vaccinations to children, and each answer is given a score from 1 to 5, with 1 being not at all confident/strongly disagree and 5 being completely confident/strongly agree. Higher numerical scores on the 5-point scale reflect higher levels of self-efficacy or confidence in personal ability to complete vaccination process actions. Study researchers will calculate the average scale based on numeric scores.

SECONDARY OUTCOMES:
Service penetration/effectiveness | Up to 12 months post intervention delivery
  Will be defined by pre and post changes in overall adolescent vaccine doses delivered across trial arms. Will present unadjusted and adjusted odds ratios accounting for multiple comparisons.
Adoption | Up to 12 months post intervention delivery
  Will be defined by pre and post changes in each pharmacy's HPV and other vaccination rates across trial arms.
Reach | Up to 12 months post intervention delivery
  Will be defined as the total number and proportion of patients who received HPV vaccination by intervention arm, overall and by patient sex, race, ethnicity, age group, insurance category, rurality, previous screening behavior, and clinic/pharmacy cluster.
Outer context/setting | Up to 24 months
  Parents will be asked to identify differences between the vaccination experience at the pharmacy compared to their child's doctor's office. Example measures: "How would you rate your pharmacy's vaccination service compared to vaccination services at your child's doctor's office?"
Inner context/setting | Up to 24 months
  In qualitative interviews, pharmacy staff will be asked about internal factors that impacted the delivery and uptake of the intervention, Example measure: "How would you rate the implementation process planning with the study team?" (Pharmacy staff; construct: Planning)
Implementation process domain | Up to 24 months
  In a qualitative interview, pharmacy staff will be asked to rate the implementation process planning with the study team.
Innovation factors/characteristics | Up to 24 months
  Pharmacy staff will be asked to compare the intervention to usual practice. Example measures: "Using the communication strategy is a better approach for delivering HPV vaccination than what I usually do."
Individuals' domain | Up to 24 months
  Assessed via qualitative interviews with pharmacy staff. Example measures: "How confident are you with counseling patients on HPV vaccine?" (pharmacy staff; construct: Self-efficacy

CONTACTS AND LOCATIONS:
Overall Officials: Parth Shah, PharmD, PhD, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (2):
- United States (2):
  - Penn State University, University Park, Pennsylvania
  - Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No